CLINICAL TRIAL: NCT03541967
Title: Study of the Hearing Performance and Comfort of a New Bone Conduction Hearing System - Comparison to the Osteo-integrated Bone Conduction Hearing Aid Mounted on a Headband: Prospective Open Multicenter Randomized Crossover Study
Brief Title: Comparison of a New Bone Conduction Hearing System to a Osteo-integrated Bone Conduction Hearing Aid on a Softband
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: overload costs
Sponsor: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MED-EL_ADHEAR_french_study1
Record Dates: First submitted 2018-05-04; First posted 2018-05-31 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Conductive Hearing Loss
Keywords: bone conduction
MeSH Terms: conditions — Hearing Loss, Conductive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ADHEAR-PONTO (Other): The ADHEAR system will be fitted to the patient who will take it at home for 15 days. Afterwards, the patient will come back to the clinical center and measurements will be done with the ADHEAR system. Then the patient will be fitted with the PONTO 3 SUPER POWER on softband and will take it at home for 15 days. Afterwards, the patient will come back to the clinical center and measurements will be done with the PONTO 3 SUPER POWER on softband.
  Interventions: Device: ADHEAR and PONTO 3 SUPER POWER on softband hearing aids
- PONTO-ADHEAR (Other): The PONTO 3 SUPER POWER on softband will be fitted to the patient who will take it at home for 15 days. Afterwards, the patient will come back to the clinical center and measurements will be done with the PONTO 3 SUPER POWER on softband. Then the patient will be fitted with the ADHEAR system and will take it at home for 15 days. Afterwards, the patient will come back to the clinical center and measurements will be done with the ADHEAR system.
  Interventions: Device: ADHEAR and PONTO 3 SUPER POWER on softband hearing aids

INTERVENTIONS:
Device: ADHEAR and PONTO 3 SUPER POWER on softband hearing aids — Device: ADHEAR non-implantable bone conduction hearing aid Comparator: PONTO 3 SUPER POWER bone conduction hearing aid with softband

SUMMARY:
Main objectives

* The first main objective is to evaluate the non-inferiority of the ADHEAR system compared to the PONTO 3 SUPERPOWER softband system in terms of average tonal gain.
* The second main objective of the study is to evaluate the superiority of the ADHEAR system compared to the PONTO 3 SUPERPOWER softband system in terms of comfort.

Secondary objectives

* Evaluate skin reactions with ADHEAR and PONTO 3 SUPER POWER on softband.
* Evaluate and compare perception in silence and noise with ADHEAR and PONTO 3 SUPER POWER on softband.
* Evaluate and compare the subjective auditory perception with ADHEAR and PONTO 3 SUPER POWER on softband.
* Evaluate the satisfaction and use of ADHEAR.

DETAILED DESCRIPTION:
Introduction

Hearing loss, or deafness, is defined by the decrease in the perception of sounds. Conductive hearing loss is characterized by damage to the outer or middle ear. Its etiologies are congenital, malformative or acquired, sequelae of infectious or inflammatory processes (chronic otitis).

They cause a defect in the transmission of the sound towards the cochlea. Conductive hearing loss can be compensated by bone conduction hearing aids or middle ear implants.

Osteo-integrated bone conduction hearing aids (Baha, Ponto) have become the standard of care for patients with conductive hearing loss when an acoustic hearing aid can't be used.

These prostheses are percutaneous but for children the implantation of the osseointegrated abutment requires that the child has developed a sufficient bone thickness. In general, surgery is not possible before the age of 5 years. [Doshi et al. 2012].

They can be mounted on headband for testing [Haute Autorité de Santé, HAS 2008] or avoid surgery especially for very young children [e.g. Hol et al. 2005, Verhagen et al. 2008, Doshi et al. 2012, Doshi and McDermott 2015]. In this case the vibration of the bone is through the skin. But these systems on headband pose problems of maintenance and pressure on the skin.

Standard headband pre-tests are recommended by HAS [HAS 2014] and the bone anchored hearing aid is a gold standard for preoperative evaluation in children. It can be used to predict the potential benefit of the implanted system [Doshi et al. 2012]. Several transcutaneous systems are developed today [Reinfelt 2015, Doshi et al. 2012, Doshi and McDermott 2015] but they also require surgery and have an age limit before implantation.

MED-EL company has developed a new bone conduction system, ADHEAR, that does not require surgery and that transmits the sound by bone vibration through the skin. This system has the advantage of not applying pressure on the skin and has no age limit.

Objective of the study:

The objective of the study is to compare the new ADHEAR bone conduction hearing aid for children with conductive hearing loss to the commonly used reference system, the osteointegrated bone conduction prosthesis.

Comparator:

The comparator is the same in all the centers and will be the PONTO 3 SUPER POWER mounted on softband.

Hypotheses

The hypotheses are that patients with the ADHEAR bone conduction hearing aid:

* do not have a mean tonal gain lower than that obtained with a PONTO 3 SUPERPOWER mounted on a softband.
* have a gain in comfort compared to a PONTO 3 SUPERPOWER mounted on a sofband

Main objectives

* The first main objective is to evaluate the non-inferiority of the ADHEAR system compared to the PONTO 3 SUPERPOWER softband system in terms of average tonal gain.
* The second main objective of the study is to evaluate the superiority of the ADHEAR system compared to the PONTO 3 SUPERPOWER softband system in terms of comfort.

Secondary objectives

* Evaluate skin reactions with ADHEAR and PONTO 3 SUPER POWER on softband.
* Evaluate and compare perception in silence and noise with ADHEAR and PONTO 3 SUPER POWER on softband.
* Evaluate and compare the subjective auditory perception with ADHEAR and PONTO 3 SUPER POWER on softband.
* To evaluate the satisfaction and use of ADHEAR.

Plan of study

It is a prospective open multicenter randomized crossover study: measures will be done on the patient at the inclusion then by randomisation a first system (ADHEAR or PONTO 3 SUPER POWER on softband) will be fit to the patient and he will take it at home for 15 days. Afterwards, the patient will come back to the clinical center and measurements will be done with the first system. Then the patient will be fitted with the second system (PONTO 3 SUPER POWER on softband or ADHEAR) and will take it at home for 15 days. Afterwards, the patient will come back to the clinical center and measurements will be done with the second system.

ELIGIBILITY:
Inclusion Criteria:

* Age: between 5 and 15 years old.
* Child for whom a bone conduction prosthesis test is indicated
* conductive hearing loss: bone conduction ≤ 10 dB Hearing Level (HL)
* Contralateral ear: air conduction ≤ 30 dB HL at 500, 1000, 2000, 3000 and 4000Hz
* No test of conductive bone conduction hearing aid with softband in the 3 months preceding the study
* No associated disorders
* Child not already fitted with a bone conduction system

Exclusion Criteria:

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-07-15 (Estimated); Primary Completion 2019-07-15 (Estimated); Study Completion 2019-07-15 (Estimated)

PRIMARY OUTCOMES:
Average tonal gain (dB) | 15 days after fitting of the system and port at home
  The threshold of free-field tonal audiometry is measured in the free field with masking of the contralateral ear with and without the auditory system. The tonal gain is defined by the difference of the tonal threshold with / without the auditory system. The average tonal gain is defined by the average of the tonal gain at frequencies 500, 1000, 2000, 3000 and 4000 Hz.
Comfort | 15 days after fitting of the system and port at home
  Perceived comfort will be measured with a visual analogue scale (VAS) of 10 cm overall comfort. The VAS will have the following anchors:
  10 = very comfortable; 8 = comfortable; 6 = comfortable enough; 4 = uncomfortable; 2 = very uncomfortable; 0 = not comfortable at all

SECONDARY OUTCOMES:
Skin reactions | 15 days after fitting of the system and port at home
  The measurement of cutaneous reactions with the auditory system will be done with a Holgers scale by the practitioner. Holgers scale:
  0 = No irritation; 1 = Slight redness; 2 = Red and slightly moist tissue; 3= Reddish and moist; 4 = Removal of hearing aid system necessary R = Removal of hearing aid system for reasons not related to skin problems
Bone conduction thresholds (dB Hearing Level (HL)) | at the inclusion and 30 days after
  The air conduction threshold conduction is measured with a headphone at 250, 500, 1000, 2000, 3000 and 4000 Hz. The variation is defined by the difference of bone conduction threshold at each frequency at the inclusion and at the end of the inclusion.
Subjective measurement of auditory perception | 15 days after fitting of the system and port at home
  The subjective auditory perception will be measured by a self-questionnaire to be completed by the parents: the Speech, Spatial, and Qualities of Hearing Scale (SSQ) for Parents [Galvin and Noble 2013]. The parents have to answer questions about specific situations for their child with and without the hearing system.
  SSQ items have VAS from 0 to 10 with integer anchors and qualitative anchors "not at all" for 0 and "perfectly" for 10.
  Scores are calculated for three subscales:
  * on speech perception: 9 VAS
  * on spatial localization: 6 VAS
  * on the quality of hearing: 8 VAS
  On each subscale the difference of score with and without the hearing system is calculated.
Measurement of satisfaction and use of ADHEAR | 15 days after fitting of the system and port at home
  The satisfaction and use of ADHEAR will be measured by a specific MED-EL self-questionnaire. Twenty questions with various qualitative answers. The analysis is descriptive for each question.
Air conduction threshold (dB HL) | at the inclusion and 30 days after
  The air conduction threshold conduction is measured with a headphone at 250, 500, 1000, 2000, 3000, 4000 and 8000 Hz. The variation is defined by the difference of air conduction threshold at each frequency at the inclusion and at the end of the inclusion.
Vocal audiometry in silence | 15 days after fitting of the system and port at home
  Measure of the speech reception threshold (i.e. the speech intensity in dB Sound Pressure Level (SPL)) for 50% (SRT50) and 100% (SRT100) of comprehension of words (list of Boorsma) in free field (with masking of the contralateral ear) with and without the auditory system. The gain (dB) is defined by the difference of SRT with/without the auditory system.
Vocal audiometry in noise | 15 days after fitting of the system and port at home
  Hirsch test in dichotic condition: signal = speech words (list of Boorsma) on the side of the auditory system ; noise = white noise at 65 dB Sound Pressure Level (SPL) in front of the patient (0°). Measure of the speech reception threshold (i.e. the speech intensity in dB SPL) for 50% (SRT50) and 100% (SRT100) of comprehension of words (list of Boorsma) in free field with and without the auditory system. The gain (dB) is defined by the difference of SRT with/without the auditory system.

IPD SHARING:
Plan to Share IPD: No